CLINICAL TRIAL: NCT05216224
Title: A Phase 2a, Randomized, Double-blind, Placebo-controlled Study to Investigate the Efficacy, Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ATI-450 vs Placebo in Patients With Moderate to Severe Hidradenitis Suppurativa (HS)
Brief Title: ATI-450 vs Placebo in Participants With Moderate to Severe Hidradenitis Suppurativa (HS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aclaris Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATI-450-HS-201
Record Dates: First submitted 2022-01-19; First posted 2022-01-31 (Actual); Results first posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis; Suppurativa; HS; Acne inversa
MeSH Terms: conditions — Hidradenitis Suppurativa; Hidradenitis

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The blinded placebo drug is packaged to match the active study drug and will be stored under the same conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ATI-450 (Experimental): ATI-450 50 milligrams (mg) oral tablet twice daily (BID)
  Interventions: Drug: ATI-450
- Placebo (Experimental): Placebo oral tablet BID
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: ATI-450 — Oral, small molecule MK2 inhibitor
  Other Names: Zunsemetinib
  Arms: ATI-450
Drug: Placebo oral tablet — Placebo tablet manufactured to match ATI-450 in appearance
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This is a Phase 2a study to investigate the efficacy, safety, tolerability, pharmacokinetics, and pharmacodynamics of ATI-450 vs placebo in patients with moderate to severe Hidradenitis Suppurativa (HS).

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and be willing to sign the Institutional Review Board (IRB)-approved participant informed consent form prior to administration of any study-related procedures.
* Participant must have stable HS.
* Total abscesses and/or nodule (AN) count of ≥5 at Baseline visit.
* HS lesions present in at least 2 distinct anatomical areas at Screening and Baseline.

Exclusion Criteria:

* Participant has a history of active skin disease other than HS that could interfere with the assessment of HS.
* Participant has an uncontrolled non-immunoinflammatory disease that may place the participant at increased risk during the study or impact the interpretation of results, e.g., previous malignancy, previous venous thromboembolism.
* Participant has experience with >2 biologics, >1 Janus kinase (JAK) inhibitor, or a combination of 1 biologic experience and 1 JAK inhibitor.
* Are currently receiving corticosteroids at doses greater than 10 mg per day of prednisone (or equivalent) or have been receiving an unstable dosing regimen of corticosteroids within 2 weeks of the Screening visit.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2021-12-29 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2023-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Aggarwal, Study Director — Aclaris Therapeutics, Inc.
Locations (20):
- United States (20):
  - Aclaris Investigational Site, Birmingham, Alabama
  - Aclaris Investigational Site, Fort Smith, Arkansas
  - Aclaris Investigational Site, Encino, California
  - Aclaris Investigational Site, San Francisco, California
  - Aclaris Investigational Site, Thousand Oaks, California
  - Aclaris Investigational Site, Boca Raton, Florida
  - Aclaris Investigational Site, Hollywood, Florida
  - Aclaris Investigational Site, Tampa, Florida
  - Aclaris Investigational Site, Marietta, Georgia
  - Aclaris Investigational Site, Sandy Springs, Georgia
  - Aclaris Investigational Site, Metairie, Louisiana
  - Aclaris Investigational Site, Fort Gratiot, Michigan
  - Aclaris Investigational Site, Charlotte, North Carolina
  - Aclaris Investigational Site, Athens, Ohio
  - Aclaris Investigational Site, Mason, Ohio
  - Aclaris Investigational Site, Hershey, Pennsylvania
  - Aclaris Investigational Site, Anderson, South Carolina
  - Aclaris Investigational Site, Nashville, Tennessee
  - Aclaris Investigational Site, Houston, Texas
  - Aclaris Investigational Site, Sugar Land, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- ATI-450: Participants received a single oral tablet of ATI-450 50 milligrams (mg) twice daily (BID) for 12 weeks.
- Placebo: Participants received a single oral tablet of Placebo BID for 12 weeks.
Period: Overall Study
Arm/Group | ATI-450 | Placebo
Started | 48 | 47
Received at Least 1 Dose of Study Drug | 48 | 47
Completed | 25 | 32
Not Completed | 23 | 15
Not completed — Adverse Event | 6 | 3
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 8 | 6
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Other than specified | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) population included all participants who have been randomized and administered at least 1 dose of study drug.
Groups:
- ATI-450: Participants received a single oral tablet of ATI-450 50 mg BID for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | ATI-450 | Placebo | Total
Number analyzed (Participants) | 48 | 47 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (9.87) | 36.6 (9.32) | 35.9 (9.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 40 | 79
  Male | 9 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 8 | 18
  Not Hispanic or Latino | 38 | 39 | 77
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 20 | 38
  White | 28 | 27 | 55
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Abscess and Inflammatory Nodule (AN) Count at Week 12
Description: AN count was the sum of number of abscess and inflammatory nodules across anatomical regions.
  The least square (LS) mean change from baseline in the count at Week 12 was estimated from the Mixed Model Repeated Measures (MMRM) model.
Time Frame: Baseline, Week 12
Population: FAS population: All participants who were randomized and administered at least 1 dose of study drug.
Measure: Least Squares Mean (90% Confidence Interval); unit: AN count
Arm/Group | ATI-450 | Placebo
Number analyzed (Participants) | 48 | 47
AN count | -2.93 [-3.99 to -1.87] | -5.94 [-7.01 to -4.87]
Statistical Analysis 1: Comparison: ATI-450 vs Placebo; Test type: Superiority; p > 0.999, MMRM — Significance level of 0.05; Fixed effect terms for treatment, study visit, treatment by visit interaction and baseline count of inflammatory abscesses and nodules as a covariate; LS Mean Difference = 3.01, 90% CI 2-sided [1.50 to 4.52]

2. Secondary Outcome: Percentage of Participants Achieving Hidradenitis Suppurativa Clinical Response (HiSCR50) at Week 12
Description: HiSCR50 Achiever was defined as a participant having a ≥50% reduction from baseline in the total abscess and inflammatory nodule count, with no increase in the number of abscesses, and no increase in the number of draining fistula counts from baseline. A participant was considered an achiever only if all 3 criteria mentioned above were fulfilled.
  Model-based estimates and 90% confidence intervals (CIs) were produced. Firth's penalized likelihood logistic regression model with fixed effects for treatment and baseline count of inflammatory abscesses and nodules was used.
Time Frame: Week 12
Population: FAS population: All participants who were randomized and administered at least 1 dose of study drug.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | ATI-450 | Placebo
Number analyzed (Participants) | 48 | 47
percentage of participants | 31.5 [21.6 to 43.4] | 51.4 [39.5 to 63.2]

3. Secondary Outcome: Change From Baseline in International Hidradenitis Suppurativa Severity Score System (IHS-4) at Week 12
Description: The IHS-4 is a validated tool used to access the HS severity and is calculated based on the clinical signs of HS: inflammatory nodules, abscesses and draining tunnels (fistulas and sinuses). The IHS-4 score = (number of nodules multiplied by 1) + (number of abscesses multiplied by 2) + (number of draining tunnels [fistulas/sinuses] multiplied by 4).
  Mild HS is a score of 3 or less, moderate HS is a score of 4-10, and severe HS is a score of 11 or higher. A decrease in score means less severity.
Time Frame: Baseline, Week 12
Population: FAS population: All participants who were randomized and administered at least 1 dose of study drug.
Measure: Least Squares Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | ATI-450 | Placebo
Number analyzed (Participants) | 48 | 47
units on a scale | -4.01 [-6.31 to -1.71] | -11.86 [-14.18 to -9.53]

4. Secondary Outcome: Percentage of Participants Achieving NRS30
Description: NRS30 Achiever was defined as participants achieving at least a 30% reduction from baseline in Patient's Global Assessment of Skin Pain (PGA-SP) and at least 1 unit reduction from baseline in PGA-SP at Week 12 among participants with baseline PGA-SP ≥3.
  Model-based estimates and 90% CIs were produced. Firth's penalized likelihood logistic regression model with fixed effects for treatment and baseline PGA-SP was used.
Time Frame: Week 12
Population: Only participants in the FAS population with a baseline NRS-PGA -SP ≥3 were evaluated for this outcome measure.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | ATI-450 | Placebo
Number analyzed (Participants) | 37 | 38
percentage of participants | 43.7 [30.9 to 57.3] | 57.5 [44.0 to 69.9]

5. Secondary Outcome: Change From Baseline in Hidradenitis Suppurativa-Physician Global Assessment (HSPGA) at Week 12
Description: In the HS-PGA scale, the Investigators rated the counts of nodules (inflammatory and non-inflammatory) abscesses and fistulas (both draining and nondraining) and assigned a participant to 1 of 6 categories ranging from clear (0) to very severe (5). A decrease in score means a better outcome.
Time Frame: Baseline, Week 12
Population: FAS population: All participants who were randomized and administered at least 1 dose of study drug.
Measure: Least Squares Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | ATI-450 | Placebo
Number analyzed (Participants) | 48 | 47
units on a scale | -0.31 [-0.48 to -0.14] | -0.73 [-0.90 to -0.55]

6. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) at Week 12
Description: The DLQI is a 10-item validated questionnaire used to assess the impact of HS disease symptoms and treatment on quality of life (QoL). It consists of questions including a single "yes/no" question and questions with possible responses of "not at all," "a little," "a lot," or "very much." These questions evaluate the impact of skin diseases on different aspects of a participant's QoL over the prior week, including symptoms and feelings, daily activities, leisure, work or school, personal relationships, and the side effects of treatment. Each question was scored using a 4-point scale ranging from 0 to 3 based on a participant's response: not at all/not relevant (0), a little (1), a lot (2) and very much (3). The total score of the DLQI ranged from 0 to 30 and was calculated by adding up the scores from each question. The higher the score, the greater the impact on a participant's QoL.
Time Frame: Baseline, Week 12
Population: FAS population: All participants who were randomized and administered at least 1 dose of study drug.
Measure: Least Squares Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | ATI-450 | Placebo
Number analyzed (Participants) | 48 | 47
units on a scale | -3.27 [-4.66 to -1.89] | -4.08 [-5.48 to -2.68]

7. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs are defined as AEs with an onset date on or after the date of first administration of study drug and before the date of last administration of study drug + 30 days. A summary of non-serious AEs and serious AEs, regardless of causality is located in Reported AEs section.
Time Frame: Baseline through Day 115
Population: Safety population: All participants randomly assigned to study drug and who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-450 | Placebo
Number analyzed (Participants) | 48 | 47
Participants | 35 | 26

8. Secondary Outcome: ATI-450 and Metabolite (CDD-2164) Concentrations
Time Frame: 2 hours postdose on Days 1, 8, and 85
Population: Pharmacokinetic (PK) population: All participants who were randomized, took at least 1 dose of study drug, and had at least 1 evaluable PK assay. Here, 'Number analyzed' = participants evaluable for specified category.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/ml)
Arm/Group | ATI-450 | Placebo
Number analyzed (Participants) | 48 | 47
Nanograms per milliliter (ng/ml)
  ATI-450 Day 1 | 144.995 (62.7707) | 0.623 (1.2728)
  ATI-450 Day 8: number analyzed (Participants) | 39 | 40
  ATI-450 Day 8 | 207.571 (98.0314) | 0.504 (1.2063)
  ATI-450 Day 85: number analyzed (Participants) | 24 | 26
  ATI-450 Day 85 | 232.110 (116.3028) | 0.250 (0.000)
  CDD-2164 Day 1 | 49.741 (26.7662) | 0.364 (0.3932)
  CDD-2164 Day 8: number analyzed (Participants) | 39 | 40
  CDD-2164 Day 8 | 63.632 (32.1682) | 0.277 (0.1231)
  CDD-2164 Day 85: number analyzed (Participants) | 24 | 26
  CDD-2164 Day 85 | 70.698 (34.0962) | 0.250 (0.000)

ADVERSE EVENTS:
Time Frame: Baseline through Day 115
Description: Safety population: All participants randomly assigned to study drug and who received at least 1 dose of study drug.
Arm/Group | ATI-450 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/48 | 1/47
Other Adverse Events (participants affected / at risk) | 23/48 | 13/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ATI-450 (N=48) | Placebo (N=47)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ATI-450 (N=48) | Placebo (N=47)
Diarrhoea (Gastrointestinal disorders) | 6 | 4
Nausea (Gastrointestinal disorders) | 2 | 3
Mouth ulceration (Gastrointestinal disorders) | 3 | 0
Fatigue (General disorders) | 3 | 0
Nasopharyngitis (Infections and infestations) | 1 | 5
COVID-19 (Infections and infestations) | 1 | 3
Blood creatine phosphokinase increased (Investigations) | 4 | 0
Dizziness (Nervous system disorders) | 8 | 0
Headache (Nervous system disorders) | 6 | 2
Acne (Skin and subcutaneous tissue disorders) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-08-04): https://cdn.clinicaltrials.gov/large-docs/24/NCT05216224/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-16): https://cdn.clinicaltrials.gov/large-docs/24/NCT05216224/SAP_001.pdf